CLINICAL TRIAL: NCT04734548
Title: A Double-Blind, Placebo-Controlled, Randomized, Phase Ib/IIa Clinical Study of ApTOLL for the Treatment of Acute Ischemic Stroke
Brief Title: Phase Ib/IIa Clinical Study of ApTOLL for the Treatment of Acute Ischemic Stroke
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: aptaTargets S.L. (Industry)
Collaborators: Ministry of Science and Innovation, Spain (Other Government); Anagram (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APRIL
Record Dates: First submitted 2021-01-28; First posted 2021-02-02 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Stroke; Acute Stroke; Ischemic Stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — TLR4 antagonist ApTOLL

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase Ib ApTOLL (Active Comparator): ApTOLL is administered intravenously in a single ascending dose pattern in four dose levels (0.025mg/kg - 0.2mg/kg). All levels include six patients.
  Interventions: Drug: ApTOLL
- Phase Ib Placebo (Placebo Comparator): Placebo is administered intravenously in a single ascending dose pattern in four dose levels (0.025mg/kg - 0.2mg/kg). All levels include two patients.
  Interventions: Other: Placebo
- Phase IIa ApTOLL (Active Comparator): ApTOLL is administered intravenously (two doses selected in Phase Ib). The two dose levels include 35 patients each one.
  Interventions: Drug: ApTOLL
- Phase IIa Placebo (Placebo Comparator): Placebo is administered intravenously in one arm which includes 49 patients.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ApTOLL — ApTOLL is a Toll-like receptor 4 (TLR4) antagonist, a receptor that is involved in innate immune responses but also responds to tissue damage, and therefore it is directly involved in a large number of diseases where the inflammatory response is involved. ApTOLL has demonstrated specific binding to human TLR4 as well as a TLR4 antagonistic effect, reducing inflammation and improving outcome after different disease models.
  Arms: Phase IIa ApTOLL; Phase Ib ApTOLL
Other: Placebo — White freeze-dried powder which is indistinguishable to ApTOLL for taste, color, texture and size.
  Arms: Phase IIa Placebo; Phase Ib Placebo

SUMMARY:
This is a prospective, multicenter, double-blind, randomized, placebo-controlled, Phase Ib/IIa clinical study to assess the administration of ApTOLL together with endovascular therapy in acute ischemic stroke patients who are candidates to receive reperfusion therapies.

DETAILED DESCRIPTION:
This is a prospective, multicenter, double-blind, randomized, placebo-controlled, Phase Ib/IIa clinical study to assess the administration of ApTOLL together with endovascular therapy in acute ischemic stroke (AIS) patients with confirmed Large Vessel Occlusion (LVO) who are candidates to receive reperfusion therapies including endovascular treatment with or without i.v. rt-PA (recombinant tissue Plasminogen Activator).

The study will be a Phase Ib/IIa trial where 2 doses selected, based on safety criteria, on Phase Ib will be administered in the following Phase IIa.The objective of the study is to evaluate if administration of ApTOLL at different doses is safe and well tolerated compared to placebo when administered with endovascular therapy (EVT), with or without i.v. rt-PA, in the AIS target population.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤90 years.
2. Informed consent obtained from subject or acceptable subject surrogate (i.e. next of kin, or legal representative).
3. A new focal disabling neurologic deficit consistent with acute cerebral ischemia.
4. Baseline NIHSS obtained prior to randomization ≥ 8 points and ≤ 25 points.
5. Pre-stroke mRS score of 0 - 2.
6. Treatable as soon as possible and at least within 6 hours of symptom onset, defined as point in time when the subject was last seen well (at baseline).
7. Patients should be candidates to receive EVT treatment with or without i.v. rt-PA.
8. Occlusion (TICI 0 or TICI 1 flow), of the terminal internal carotid artery (TICA), M1 or M2 segments of the middle cerebral artery, suitable for mechanical embolectomy, confirmed on Computed Tomography Angiography.
9. The following imaging criteria should also be met on admission neuroimaging:

   1. MRI criterion: volume of DWI (Diffusion-weighted Imaging) restriction ≥5 mL and ≤70 mL OR
   2. CT criterion: Alberta Stroke program early CT score (ASPECTS) 6 to 10 on baseline CT AND infarct core determined on admission CTPerfusion by Cerebral Blood Flow<30%: ≥5 mL and ≤70 mL.
10. The subject has an indication and is planned to receive endovascular treatment of stroke according to the European Stroke Organization Guidelines.

Exclusion Criteria:

1. Subject has suffered a stroke in the past 1 year.
2. Occlusion (TICI 0 or TICI 1 flow) of the basilar or vertebral or posterior or anterior cerebral arteries.
3. Clinical symptoms suggestive of bilateral stroke or stroke in multiple territories.
4. Known hemorrhagic diathesis, coagulation factor deficiency, or oral anticoagulant therapy with INR (international normalized ratio)>3.0.
5. Baseline platelet count <50,000/μL.
6. Baseline blood glucose of <50 mg/dL or >400 mg/dL.
7. Severe, sustained hypertension (systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg).
8. Serious, advanced, or terminal illness with anticipated life expectancy of less than 1 year.
9. Subjects with identifiable intracranial tumors.
10. History of life-threatening allergy (more than rash) to contrast medium.
11. Known renal insufficiency with creatinine ≥3 mg/dL or Glomerular Filtration Rate (GFR) <30 mL/min.
12. Cerebral vasculitis.
13. Evidence of active systemic infection.
14. Known current use of cocaine at time of treatment.
15. Patient participating in a study involving an investigational drug or device that would impact this study.
16. Patients that are unlikely to be available for a 90-day follow-up (e.g. no fixed home address, visitor from overseas).
17. Female who is pregnant or lactating or has a positive pregnancy test at time of admission.
18. CT or MRI evidence of hemorrhage (the presence of microbleeds is allowed).
19. Significant mass effect with midline shift.
20. Suspicion of aortic dissection presumed septic embolus, or suspicion of bacterial endocarditis.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Safety of ApTOLL | From dosing to follow-up (day 90 after dosing)
  To assess if ApTOLL is safe when combined with EVT therapy as determined by:
  1. Death.
  2. Adverse events that occur during the study.
  3. Physical examination.
  4. Laboratory tests.
  5. Recurrent stroke.
  6. Symptomatic intracranial hemorrhage (sICH).

SECONDARY OUTCOMES:
Mean infarct volume | 72 hours
  Magnetic Resonance Image
Effect in inflammatory response | Predose and up to 72 hours post-dose
  Proinflammatory markers in blood between study groups
Early clinical course | 72 hours post-dose
  NIHSS (National institute of Health Stroke Scale). The maximum possible score is 42, with the minimum score being a 0 (the higher the score, the more impaired a stroke patient is)
Long-term outcome | Day 90 post-dose
  mRS (modified Ranking Score). Coded from 0 (no symptoms at all) through 5 (severe disability) 6 (death).

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ribó, MD, PhD, Study Director — aptaTargets S.L.; Macarena Hernández, PhD, Study Director — aptaTargets S.L.
Locations (16):
- France (3):
  - Centre Hospitalier Régional Universitaire de Lille, Lille
  - Foundation Adolphe de Rothschild, Paris
  - Centre Hospitalier Universitaire de Toulouse, Toulouse
- Universitätsklinikum Essen, Essen, Germany
- Spain (12):
  - Hospital Universitario A Coruña, A Coruña
  - Hospital Universitario Central de Asturias, Asturias
  - Hospital Bellvitge, Barcelona
  - Hospital Germans Trias i Pujol, Barcelona
  - Hospital Universitario Vall d´Hebron, Barcelona
  - Hospital Universitario de Gerona Dr. Josep Trueta, Girona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Virgen del Rocío, Seville
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital Clínico Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No
All results obtained in this study will be published.

REFERENCES:
- [Background] Hernandez-Jimenez M, Martin-Vilchez S, Ochoa D, Mejia-Abril G, Roman M, Camargo-Mamani P, Luquero-Bueno S, Jilma B, Moro MA, Fernandez G, Pineiro D, Ribo M, Gonzalez VM, Lizasoain I, Abad-Santos F. First-in-human phase I clinical trial of a TLR4-binding DNA aptamer, ApTOLL: Safety and pharmacokinetics in healthy volunteers. Mol Ther Nucleic Acids. 2022 Mar 9;28:124-135. doi: 10.1016/j.omtn.2022.03.005. eCollection 2022 Jun 14. PMID 35402075
- [Derived] Hernandez-Jimenez M, Abad-Santos F, Cotgreave I, Gallego J, Jilma B, Flores A, Jovin TG, Vivancos J, Hernandez-Perez M, Molina CA, Montaner J, Casariego J, Dalsgaard M, Liebeskind DS, Cobo E, Castellanos M, Portela PC, Masjuan J, Moniche F, Tembl JI, Terceno Izaga M, Arenillas JF, Callejas P, Olivot JM, Calviere L, Henon H, Mazighi M, Pineiro D, Pugliese M, Gonzalez VM, Moro MA, Garcia-Tornel A, Lizasoain I, Ribo M. Safety and Efficacy of ApTOLL in Patients With Ischemic Stroke Undergoing Endovascular Treatment: A Phase 1/2 Randomized Clinical Trial. JAMA Neurol. 2023 Aug 1;80(8):779-788. doi: 10.1001/jamaneurol.2023.1660. PMID 37338893
- [Derived] Hernandez-Jimenez M, Abad-Santos F, Cotgreave I, Gallego J, Jilma B, Flores A, Jovin TG, Vivancos J, Molina CA, Montaner J, Casariego J, Dalsgaard M, Hernandez-Perez M, Liebeskind DS, Cobo E, Ribo M. APRIL: A double-blind, placebo-controlled, randomized, Phase Ib/IIa clinical study of ApTOLL for the treatment of acute ischemic stroke. Front Neurol. 2023 Feb 24;14:1127585. doi: 10.3389/fneur.2023.1127585. eCollection 2023. PMID 36908619
- [Derived] Duran-Laforet V, Pena-Martinez C, Garcia-Culebras A, Alzamora L, Moro MA, Lizasoain I. Pathophysiological and pharmacological relevance of TLR4 in peripheral immune cells after stroke. Pharmacol Ther. 2021 Dec;228:107933. doi: 10.1016/j.pharmthera.2021.107933. Epub 2021 Jun 24. PMID 34174279
- See also: Biotechnology company specialized in therapeutic aptamers — http://aptatargets.com